CLINICAL TRIAL: NCT01216176
Title: A Phase I Pharmacokinetic and Randomized Phase II Trial of Neoadjuvant Treatment With Anastrozole Plus AZD0530 in Postmenopausal Patients With Hormone Receptor Positive Breast Cancer
Brief Title: A Pharmacokinetic and Randomized Trial of Neoadjuvant Treatment With Anastrozole Plus AZD0530 in Postmenopausal Patients With Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joyce Marie Slingerland, MD (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Joyce Marie Slingerland, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080325; SCCC-2008002 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Postmenopausal; Metastatic Phase I ONLY; AZD0530 (saracatinib); Anastrozole; Phase I for metastatic disease; Phase II for newly diagnosed breast cancer; Pharmacokinetic; PK; Hormone Receptor; Estrogen Receptor; Progesterone Receptor; ER+; PR+; HER negative; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; saracatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 - Cohort A (Experimental): Dual treatment with 1 mg anastrozole orally once daily together with AZD0530 (saracatinib) 175 mg orally once daily, or as specified per protocol, until disease progression for treatment of metastatic breast cancer
  Interventions: Drug: Anastrozole; Drug: AZD0530 (saracatinib)
- Phase 2 - Cohort B [Anastrozole + AZD0530] (Active Comparator): Dual treatment with 1 mg anastrozole orally once daily together with AZD0530 (saracatinib) 175 mg orally once daily, or as specified per protocol, until disease progression or 4-6 months of treatment completed.
  Interventions: Drug: Anastrozole; Drug: AZD0530 (saracatinib)
- Phase 2 - Cohort B [Anastrozole + Placebo] (Placebo Comparator): Dual treatment with 1 mg anastrozole orally once daily together with Placebo orally once daily, or as specified per protocol, until disease progression or4-6 months of treatment completed.
  Interventions: Drug: Anastrozole; Drug: Placebo

INTERVENTIONS:
Drug: Anastrozole
Drug: AZD0530 (saracatinib)
  Arms: Phase 1 - Cohort A; Phase 2 - Cohort B [Anastrozole + AZD0530]
Drug: Placebo
  Arms: Phase 2 - Cohort B [Anastrozole + Placebo]

SUMMARY:
The investigators propose to conduct a Phase I/randomized Phase II study design in order to test the tolerability and efficacy of AZD0530 (also called saracatinib) when used together with anastrozole in therapy for ER+ and/or PR+, postmenopausal breast cancer. The Phase I pharmacokinetic (PK) cohort of the study (cohort A) in postmenopausal women with metastatic breast cancer 2008-2009 showed initial safety,tolerability and good bioavailability of both drugs and determined the doses for use in the ongoing Phase II trial. In the randomized Phase II cohort of the study (cohort B), postmenopausal women with newly diagnosed, previously untreated ER+, HER2 negative breast cancer that is at least 2 cm or more in diameter by clinical exam or radiology will be randomized to either neoadjuvant treatment with anastrozole plus placebo, or anastrozole in combination with AZD0530 (saracatinib). The Phase II cohort will permit extended assays of tolerability, initial estimates of efficacy, and the investigation of molecular predictors of drug efficacy.

ELIGIBILITY:
Inclusion Criteria - Phase 1 (Cohort A):

* Female patient ≥ 18 years
* Patient must be postmenopausal, verified by 1 of the following:

  * Bilateral surgical oophorectomy
  * No spontaneous menses > 1 year
  * No menses for < 1 year with FSH and estradiol levels in postmenopausal range. If a study subject under the age of 60 reports prior surgery in which the ovaries were removed and if the operative report cannot be obtained to confirm bilateral salpingo-oophorectomy, the subject will have serum estradiol, LH and FSH drawn to confirm menopausal status prior to study entry
* Postmenopausal women with primary invasive breast cancer, histologically confirmed by core needle (or incisional biopsy), whose tumors are estrogen (ER) and/or progesterone (PgR) positive. Estrogen- and/or progesterone-receptor positive disease based on 10% or more nuclear staining of the invasive component of the tumor
* Stage IV disease (as defined by the AJCC Staging Manual, 6th Edition, 2002); or locally relapsed, unresectable disease
* Measurable or evaluable disease according to RECIST criteria (see appendix VII)
* Both HER2-positive and HER2-negative disease (as defined by IHC or by fluorescence in situ hybridization [FISH]). HER2+ must have had prior treatment with trastuzumab and/or lapatinib.
* ECOG performance status 0-2 (see appendix VI)
* Patients are suitable candidates for treatment with anastrozole (patients may have had any prior endocrine therapy or prior chemotherapy for treatment of their disease, either as adjuvant therapy, or as treatment for advanced disease). There is no restriction on the number of prior regimens in the phase I cohort A.
* Patient is accessible and willing to comply with treatment and follow-up
* Patient is willing to provide written informed consent prior to the performance of any study-related procedures
* Required laboratory values

  * Absolute neutrophil count ≥ to 1.5 x 10^9/L
  * Hemoglobin ≥ to 9.0 g/dL
  * Platelet count ≥ to 100 x 10^9/L
  * Creatinine ≤ 1.5 mg/dL
  * Total bilirubin ≤ 1.0 x upper limit of normal (ULN)
  * Alkaline phosphatase and AST/ALT within protocol parameters. In determining eligibility, the more abnormal of the two values (AST or ALT) should be used.

Inclusion Criteria - Phase 2 (Cohort B):

* Female patient ≥ 18 years
* Patient must be postmenopausal, verified by 1 of the following:

  * Bilateral surgical oophorectomy
  * No spontaneous menses ≥ 1 year
  * No menses for < 1 year with FSH and estradiol levels in postmenopausal range. If a study subject under the age of 60 reports prior surgery in which the ovaries were removed and if the operative report cannot be obtained to confirm bilateral salpingo-oophorectomy, the subject will have serum estradiol, LH and FSH drawn to confirm menopausal status prior to study entry
* Postmenopausal women with primary invasive breast cancer, histologically confirmed by core needle (or incisional biopsy), whose tumors are estrogen (ER) and/or progesterone (PgR) positive. Estrogen- and/or progesterone-receptor positive disease based on 10% or more nuclear staining of the invasive component of the tumor. Patients may have bilateral or multifocal invasive breast cancers. The patient may have concurrent DCIS in either breast but the DCIS will not be measured as part of the study endpoints.
* Tumor size ≥ 2 cm
* Tumor measurable either by clinical examination, mammography, MRI, or ultrasound
* HER2-negative disease (as defined by fluorescence in situ hybridization [FISH] or by IHC)
* ECOG performance status 0-1 (see Appendix VI)
* Patient is accessible and willing to comply with treatment and follow-up
* Patient is willing to provide written informed consent prior to the performance of any study-related procedures
* Required laboratory values

  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 70 x 10^9/L
  * Creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase and AST/ALT ≤ 1.5 x upper limit of normal (ULN)

Exclusion Criteria - Phase 1 (Cohort A):

* Concurrent therapy with any other non-protocol anti-cancer therapy

  * Any agent with estrogenic or putatively estrogenic properties, including herbal preparations, must be stopped at least one week prior to registration.
  * Ongoing, chronic administration of bisphosphonate therapy is allowed so long as such treatment was ongoing at the time of study entry.
* Current therapy with hormone replacement therapy, or any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (agents must be stopped prior to randomization)
* Presence of neuropathy ≥ grade 2 (NCI-CTC version 3.0) at baseline
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease (e.g., hypertension [BP > 150/100], history of myocardial infarction or stroke within 6 months, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Active, uncontrolled infection requiring parenteral antimicrobials
* A history of a severe hypersensitivity reaction to anastrozole, or AZD0530 or their excipients
* Evidence of bleeding diathesis or coagulopathy.
* Resting EKG with measurable QTc interval of >480msec at 2 or more time points within a 24 hr period.
* Since AZD0530 is a substrate and inhibitor of CYP3A4, patients requiring medication with drugs listed in Appendix XI should be excluded from study.
* Any evidence of severe or uncontrolled systemic medical or psychiatric conditions (e.g. Severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]) or current unstable or uncompensated respiratory or cardiac conditions which make it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
* Evidence of underlying pulmonary dysfunction as evidenced by oxygen saturation <90% by pulse oximetry, interstitial pulmonary infiltrates on high resolution CT scan prior to study entry and/or symptomatic pulmonary (pleural or parenchymal) metastasis.

Exclusion Criteria - Phase 2 (Cohort B):

* Prior chemotherapy, endocrine therapy or radiotherapy for the presenting breast cancer. Prior incidence and treatment of contralateral invasive or non-invasive breast cancer is not an exclusion criterion.
* Inflammatory breast cancer, clinically defined as the presence of erythema or induration involving one-third or more of the breast, or pathologically defined as dermal lymphatic invasion
* Prior excisional biopsy or complete resection of the primary invasive tumor (prior sentinel node biopsy allowed)
* Prior ipsilateral radiation therapy for invasive or non-invasive breast cancer
* Distant metastasis is an exclusion criterion - Isolated ipsilateral supraclavicular node involvement and/or direct invasion of the primary tumor into skin is allowed
* Concurrent therapy with any other non-protocol anti-cancer therapy
* Any agent with estrogenic or putatively estrogenic properties, including herbal preparations, must be stopped at least one week prior to registration
* Current therapy with hormone replacement therapy, or any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (agents must be stopped for one week prior to randomization)
* Presence of neuropathy ≥ grade 2 (NCI-CTC AE version 3.0) at baseline
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease (e.g. history of myocardial infarction or stroke within 6 months, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Active, uncontrolled infection requiring parenteral antimicrobials
* A history of a severe hypersensitivity reaction to anastrozole, or AZD0530 (saracatinib) or their excipients
* Evidence of bleeding diathesis or coagulopathy
* Resting EKG with measurable QTc interval of >480msec at 2 or more time points within a 24 hr period.
* AZD0530 (saracatinib) is a substrate and inhibitor of CYP3A4. Since concurrent administration of AZD0530 with other CYP3A4 substrates has been shown to be well tolerated, continuation or initiation of medically indicated drugs that are substrates of CYP3A4 is permitted at MD discretion. Drugs listed in Appendix X that are known to strongly induce or inhibit CYP3A4 activity should be discontinued prior to study entry and should not be initiated during protocol treatment.
* Any evidence of severe or uncontrolled systemic psychiatric or medical conditions (eg. Severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]) or current unstable or uncompensated respiratory or cardiac conditions which make it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
* Evidence of underlying pulmonary dysfunction as evidenced by oxygen saturation <90% by pulse oximetry prior to study entry and/or symptomatic pulmonary (pleural or parenchymal) disease.
* Subjects unwilling or unable to undergo breast MRI as required by protocol will be excluded from study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-10-21 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Slingerland, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of Miami, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the Phase 1 cohort, all 12/12 planned subjects were accrued. Of the planned 60 subjects for Phase 2, 59 subjects were accrued. One was removed from study within a few days ( MD discretion) and is not included in subsequent analysis.
Groups:
- Phase 1 - Cohort A: Dual treatment with 1 mg anastrozole orally once daily together with AZD0530 175 mg orally once daily, or as specified per protocol, until disease progression for treatment of metastatic breast cancer
  Anastrozole
  AZD0530
- Phase 2 - Cohort B [Anastrozole + AZD0530]: Dual treatment with 1 mg anastrozole orally once daily together with AZD0530 175 mg orally once daily, or as specified per protocol, until disease progression or 4-6 months of treatment completed.
  Anastrozole
  AZD0530
- Phase 2 - Cohort B [Anastrozole + Placebo]: Dual treatment with 1 mg anastrozole orally once daily together with Placebo orally once daily, or as specified per protocol, until disease progression or4-6 months of treatment completed.
  Anastrozole
  Placebo
Period: Overall Study
Arm/Group | Phase 1 - Cohort A | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Started | 12 | 39 | 20
Completed | 12 | 31 | 19
Not Completed | 0 | 8 | 1
Not completed — Adverse Event | 0 | 8 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Cohort A | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo] | Total
Number analyzed (Participants) | 12 | 39 | 20 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 28 | 16 | 55
  >=65 years | 1 | 11 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 39 | 20 | 71
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic white | 9 | 9 | 1 | 19
  Race/Ethnicity: Non-Hispanic black or African America | 0 | 4 | 5 | 9
  Race/Ethnicity: Hispanic | 3 | 24 | 12 | 39
  Race/Ethnicity: Asian | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase I Cohort A: Maximum Tolerated AZD0530 Daily Dose Used in Combination With Daily Oral Anastrozole
Description: To identify a well tolerated dose of AZD0530 (saracatinib) that can be used together with anastrozole in the Phase 2 trial with tolerable toxicity and PK, subjects were followed as AEs recorded and evaluated and drug concentrations were in the therapeutic range.
Time Frame: Cycle 1: Days 1 - 28
Population: All participants enrolled to phase 1.
Measure: Number; unit: mg/day oral dose
Arm/Group | Phase 1 - Cohort A
Number analyzed (Participants) | 12
mg/day oral dose
  anastrozole | 1
  saracatinib | 175

2. Primary Outcome: Phase II - Cohort B: Compare Treatment Groups (AZD0530 + Anastrozole Versus Anastrozole With Placebo) With Respect to Clinical Response
Description: Clinical response is defined as percentage change in tumor size calculated from bi-dimensional clinical tumor measurement at diagnosis and on completion of neoadjuvant treatment. The mean reduction in tumor size ( +/-SD) will be derived form the change in largest tumor dimension ( RECIST) and by calculated tumor volume
Time Frame: Baseline, cycle 6
Population: Of 59 subjects, 2 (one/arm)tumors were not palpable at baseline; 1 was removed at MD discretion; 8 removed due to AEs . 48 (30+18) completed 4 mo of therapy and were evaluable for clinical response. Subjects completing 4 months were permitted to go tor surgery. At 24 weeks 19 dual and 16 monotherapy remained evaluable for clinical tumor size.
Measure: Mean (Standard Deviation); unit: percentage of tumor volume change
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 19 | 16
percentage of tumor volume change
  Max clinical diameter % change | -61.5 (22.5) | -62.3 (25)
  Clinical tumor volume% change | -87.9 (22.6) | -90.7 (11.8)

3. Secondary Outcome: Phase I - Cohort A: Plasma Concentrations of AZD0530 (Saracatinib) and Anastrozole
Description: Summarized as mean plasma concentrations (ng/ml) of each drug (AZD0530 (saracatinib) and Anastrozole) after exposure to dual therapy.
Time Frame: 0 hrs, 6 hrs, 12 hrs, 24hrs, 48 hrs, 72 hrs, 8 days, 15 days, 22 days after first dose of AZD0530
Population: Day 21 - 1 missing sample.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Phase 1 - Cohort A: Dual treatment with 1 mg anastrozole orally once daily given for 7 days followed by anastrozole 1 mg orally once daily together with AZD0530 175 mg orally once daily, or as specified per protocol, until disease progression for treatment of metastatic breast cancer.
  Anastrozole
  AZD0530
Arm/Group | Phase 1 - Cohort A
Number analyzed (Participants) | 12
ng/ml
  AZD0530 - Cycle 1: 0 hrs | 0 (0)
  AZD0530 - Cycle 1: 6 hrs | 127.47 (57.12)
  AZD0530 - Cycle 1: 12 hrs | 79.1 (33.42)
  AZD0530 - Cycle 1: 24 hrs | 46.17 (24.86)
  AZD0530 - Cycle 1: 48 hrs | 91.33 (39.60)
  AZD0530 - Cycle 1: 72 hrs | 125.49 (52.63)
  AZD0530 - Day 8 | 232.23 (91.54)
  AZD0530 - Day 15 | 213.52 (84.13)
  AZD0530 - Day 22: number analyzed (Participants) | 11
  AZD0530 - Day 22 | 271.97 (144.07)
  Anastrozole - Day 1: 0 hrs | 26.35 (11.55)
  Anastrozole - Day 1: 6 hrs | 38.2 (26.88)
  Anastrozole - Day 1: 12 hrs | 33.45 (22.13)
  Anastrozole - (24 hrs) | 29.33 (21.49)
  Anastrozole - (48 hrs) | 32.81 (25.15)
  Anastrozole - (72 hrs) | 34.08 (20.01)
  Anastrozole - Day 8 | 51.00 (22.69)
  Anastrozole - Day 15 | 46.75 (28.07)
  Anastrozole - Day 22 | 47.33 (25.15)

4. Secondary Outcome: Phase 1-Cohort A: Peak Concentration of Each Study Drug ( AZD0530 (Saracatinib) and Anastrozole)
Description: Summarized as the geometric means and standard deviations for the corresponding for peak plasma concentration of each study drug ( AZD0530 (saracatinib) and anastrozole) after exposure
Time Frame: 0 hrs, 6 hrs, 12 hrs, 24hrs, 48 hrs, 72 hrs, 7 days, 14 days, 21 days after first dose of AZD0530
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | Phase 1 - Cohort A
Number analyzed (Participants) | 12
ng/ml
  AZD0530 (saracatinib) ng/ml | 271.97 (144.07)
  anastrozole ng/ml | 47.33 (25.15)

5. Secondary Outcome: Phase II Cohort B: Change in Tumor Size by Comparison of Serial MRI
Description: MRI will be used to compare tumor size at baseline and at 10 weeks. MRI will also be used to compare tumor size at baseline and after completion of 6 months of study medication or disease progression.
Time Frame: Baseline to 10 weeks;and baseline to 6 months
Population: Of 59 subjects, 1 was removed at MD discretion; 8 removed due to AEs. Of the remaining 50 (31 dual + 19 mono), all had MRI at 10 weeks. 3 dual and 1 mono had disease progression and no further MRIs. 7 out of 28 (dual) & 2 out 18 (mono) completing 4 months, had end of study MRI at wk 18; 21 ( dual) and 16 (mono) had a final MRI at 24 weeks .
Measure: Mean (Standard Deviation); unit: percentage of tumor volume change
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 31 | 19
percentage of tumor volume change
  MRI RECIST % change 10 weeks | -26.9 (30.4) | -15.9 (19.6)
  MRI tumor volume % change 10 weeks | -46.4 (43.1) | -35.0 (31.7)
  MRI RECIST % change 6 months: number analyzed (Participants) | 21 | 16
  MRI RECIST % change 6 months | -44.6 (34.1) | -22.5 (27.1)
  MRI tumor volume % change 6 months: number analyzed (Participants) | 21 | 16
  MRI tumor volume % change 6 months | -70.7 (29.5) | -43.2 (50.9)

6. Secondary Outcome: Phase II - Cohort B: Number of Participants With Pathologic Complete Response (pCR)
Description: A pathologic complete response will be defined as the absence of viable tumor cells in the resected specimen, as determined by standard histologic examination. All specimens will be reviewed by a central pathologist to determine pathologic response.
Time Frame: At completion of 4-6 cycles of therapy or after disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 31 | 19
Participants | 0 | 0

7. Secondary Outcome: Phase II - Cohort B: The Number of Participants Achieving Clinical Benefit Defined as Complete Response (CR), or Partial Response (PR) or Stable Disease (SD)
Description: Based on physician measurement of tumor size and by MRI measurements of tumor volume using RECIST criteria
Time Frame: At the end of neoadjuvant therapy
Population: 8 patients were removed from the study due to adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 23 | 19
Participants
  Complete Response | 0 | 0
  Partial Response | 16 | 17
  Stable Disease | 0 | 0
  Disease Progression | 7 | 2

8. Secondary Outcome: Phase II - Cohort B: To Report the Pharmacokinetics (Mean Blood Levels of Drug) of AZD0530 (Saracatinib) and Anastrozole
Description: Blood draws at protocol-specified timepoints to determine mean blood levels of drug for each of AZD0530 and Anastrozole.
Time Frame: Day 28, 56, 84
Population: PK assays of AZD0530 could not be completed for all participants due to technical problems with the assay protocol
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 39 | 19
ng/ml
  Anastrozole - Day 28: number analyzed (Participants) | 37 | 18
  Anastrozole - Day 28 | 52.7 (22.3) | 37.4 (10.4)
  Anastrozole - Day 56: number analyzed (Participants) | 33 | 19
  Anastrozole - Day 56 | 49.9 (21) | 37.6 (12.3)
  Anastrozole - Day 84: number analyzed (Participants) | 31 | 18
  Anastrozole - Day 84 | 48.3 (17.2) | 39.5 (11.7)
  AZD0530 - Day 28: number analyzed (Participants) | 7 | 0
  AZD0530 - Day 28 | 264.6 (96.8) |
  AZD0530 - Day 56: number analyzed (Participants) | 5 | 0
  AZD0530 - Day 56 | 286.4 (65.9) |
  AZD0530 - Day 84: number analyzed (Participants) | 5 | 0
  AZD0530 - Day 84 | 258.6 (100.9) |

9. Secondary Outcome: Phase II - Cohort B: Treatment Emergent Adverse Events Associated With AZD0530 (Saracatinib) Given With Anastrozole and of Anastrozole Given With Placebo
Description: Cinically significant AEs defined as clinically significant changes in the patient's symptoms, physical examination and clinical laboratory results are reported as toxicity for AZD0530 (saracatinib) given with anastrozole and for anastrozole given with placebo
Time Frame: From day 1 of treatment until a maximum of 6 months of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
Number analyzed (Participants) | 31 | 19
Participants
  Anemia | 7 | 1
  Neutropenia | 4 | 1
  Thrombocytopenia | 3 | 0
  Fatigue | 10 | 3
  Rash | 24 | 3
  Alopecia | 17 | 2
  Hot Flashes | 18 | 7
  Anorexia | 8 | 1
  Diarrhea | 23 | 6
  Alanine aminotransferase increased | 19 | 3
  Alkaline phosphatase increased | 11 | 0
  Aspartate aminotransferase increased | 20 | 1
  Creatinine increased | 3 | 1
  Hyperbilirubinemia | 3 | 0
  Flu-like syndrome | 9 | 1
  Upper Respiratory Infection | 14 | 2
  Urinary Tract Infection | 13 | 1

ADVERSE EVENTS:
Time Frame: 8 months. Adverse event data were collected from study entry until subjects were taken off therapy
Arm/Group | Phase 1 - Cohort A | Phase 2 - Cohort B [Anastrozole + AZD0530] | Phase 2 - Cohort B [Anastrozole + Placebo]
All-Cause Mortality (participants affected / at risk) | 2/12 | 0/39 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/12 | 5/39 | 1/20
Other Adverse Events (participants affected / at risk) | 12/12 | 39/39 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Cohort A (N=12) | Phase 2 - Cohort B [Anastrozole + AZD0530] (N=39) | Phase 2 - Cohort B [Anastrozole + Placebo] (N=20)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Brain hemorrhage complicating CNS metastasis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — One patient had a MI and congestive heart failure felt to be unrelated to study drug
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — The subject with MI also had congestive heart failure unrelated to study drug
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — This diabetic patient developed a drug related rash but was admitted to hospital because the steroid treatment precipitated hyperglycemia and admission to hospital
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Cohort A (N=12) | Phase 2 - Cohort B [Anastrozole + AZD0530] (N=39) | Phase 2 - Cohort B [Anastrozole + Placebo] (N=20)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 7 (7) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 8 (8) | 7 (7) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0)
Fatigue (General disorders) | 5 (5) | 10 (10) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 24 (24) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 17 (17) | 2 (2)
Hot flashes (Endocrine disorders) | 3 (3) | 18 (18) | 7 (7)
Anorexia (Gastrointestinal disorders) | 4 (4) | 8 (8) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 23 (23) | 6 (6)
Alanine aminotransferase increased (Hepatobiliary disorders) | 4 (4) | 19 (19) | 3 (3)
Alkaline phosphatase increased (Hepatobiliary disorders) | 5 (5) | 11 (11) | 0 (0)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 6 (6) | 20 (20) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
Flu-like syndrome (General disorders) | 1 (1) | 9 (9) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 14 (14) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 13 (13) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 3 (3) | 0 (0)
Insomnia (General disorders) | 1 (1) | 3 (3) | 0 (0)
Sweating (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Investigations) | 0 (0) | 3 (3) | 6 (6)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
Hyponatremia (Investigations) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (11) | 4 (4)
Joint Function (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 13 (13) | 7 (7)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Conjuntivitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 0 (0)
Vaginal infection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT01216176/Prot_SAP_000.pdf